CLINICAL TRIAL: NCT03238495
Title: Randomized Trial of Neo-adjuvant Chemotherapy With or Without Metformin for HER2 Positive Operable Breast Cancer
Acronym: HERMET
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qamar Khan (Other)
Responsible Party: Sponsor-Investigator, Qamar Khan, Associate Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00140673
Record Dates: First submitted 2017-07-31; First posted 2017-08-03 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: HER2-positive Breast Cancer
Keywords: Operable breast cancer; Neo-adjuvant chemotherapy
MeSH Terms: interventions — Docetaxel; Carboplatin; Trastuzumab; pertuzumab; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chemotherapy Only (Active Comparator): Taxotere, Carboplatin, Herceptin + Pertuzumab (TCH+P)
  Interventions: Drug: Taxotere, Carboplatin, Herceptin + Pertuzumab
- Chemotherapy plus Metformin (Experimental): TCH+P plus metformin
  Interventions: Drug: Taxotere, Carboplatin, Herceptin + Pertuzumab; Drug: Metformin

INTERVENTIONS:
Drug: Taxotere, Carboplatin, Herceptin + Pertuzumab — TCH+P chemotherapy every 3 weeks for 6 cycles: Taxotere 75mg/m2, Carboplatin AUC 6, Herceptin 6mg/kg (first cycle loading dose of 8mg/kg), Pertuzumab 420mg (first cycle loading does of 840mg)
Drug: Metformin — TCH+P chemotherapy every 3 weeks for 6 cycles. Metformin 850 mg daily during the first cycle, then 850 mg twice daily for the remaining 5 cycles.
  Arms: Chemotherapy plus Metformin

SUMMARY:
The primary objective of this study is to determine the efficacy of metformin as a repurposed agent in human epidermal growth factor receptor 2 (HER2) positive breast cancer when added to standard neo-adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0-1.
* Unilateral or bilateral primary carcinoma of the breast, confirmed histologically by needle core biopsy. Fine-needle aspiration is not sufficient. Incisional/excisional biopsy is not allowed. In case of bilateral cancer, the investigator has to decide prospectively which side will be evaluated for the primary endpoint.
* Study participants must be cT1c - cT4a-d, any node (N), no metastases (M0). Any tumor (T) is allowed if node positive (biopsy proven and HER2 positive) including no primary invasive cancer or only ductal carcinoma in situ (DCIS). Metastatic workup is not required.
* Breast tumor must be >1.5 cm in maximum diameter by clinical or any radiologic measurement, if node negative. If node is positive by biopsy, study participant will be eligible regardless of the size of the breast primary. In case of inflammatory breast cancer, the extent of inflammation/erythema can be used as measurable lesion.
* Multifocal or multicentric breast cancer is allowed if all the lesions are biopsied and are HER2 positive. Largest lesion will be assigned the target lesion.
* Must be HER2-positive in primary breast tumor or lymph node by the ASCO/CAP guidelines 2013: http://www.asco.org/guidelines/her2
* Ejection fraction (EF) greater than 50% by MUGA or ECHO within 4 weeks prior to first dose of study treatment.
* No prior cancer chemotherapy allowed.
* Adequate organ and marrow function as defined below, unless deemed non-clinically significant and approved by the Principal Investigator:

  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcl
  * total bilirubin within normal institutional limits
  * AST(SGOT) ≤ 2.5 X institutional upper limit of normal
  * ALT(SPGT) ≤ 2.5 X institutional upper limit of normal
  * ALK Phos ≤ 2.5 X institutional upper limit of normal
  * Creatinine clearance > 50mL/min
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy.
* Negative pregnancy test within 14 days prior to randomization

Exclusion Criteria:

* Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the study participant or the quality of the study data.
* Current or anticipated use of other investigational agents.
* Prior chemotherapy for any malignancy.
* Prior radiation therapy for breast cancer
* Previous malignant disease being disease-free for less than 5 years (except carcinoma in situ (CIS) of the cervix and non-melanoma skin cancer).
* Patients with diabetes on metformin. Patients with diabetes and not on metformin will be eligible if it is deemed safe after consultation with the patient physician managing diabetes.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to metformin or other agents used in study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-08-15 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) | Up to 6 weeks after last chemotherapy treatment
  pCR at surgery

CONTACTS AND LOCATIONS:
Overall Officials: Qamar Khan, MD, Principal Investigator — University of Kansas Medical Center
Locations (6):
- United States (6):
  - The University of Kansas Cancer Center, West Clinic, Kansas City, Kansas
  - The University of Kansas Cancer Center, Westwood Campus, Kansas City, Kansas
  - The University of Kansas Cancer Center, Overland Park Clinic, Overland Park, Kansas
  - The University of Kansas Cancer Center, South Clinic, Kansas City, Missouri
  - The University of Kansas Cancer Center, North Clinic, Kansas City, Missouri
  - The University of Kansas Cancer Center, Lee's Summit Clinic, Lee's Summit, Missouri

IPD SHARING:
Plan to Share IPD: No